CLINICAL TRIAL: NCT03323333
Title: Psychosocial Intervention Pilot for Partners in BRCA Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-0907
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Behavioral: psychosocial counseling

INTERVENTIONS:
Behavioral: psychosocial counseling — A problem-solving and psychosocial skill-building intervention.

SUMMARY:
A brief psychosocial intervention for partners of women affected by or at risk for breast cancer and harboring BRCA genetic alterations.

ELIGIBILITY:
Inclusion Criteria:

* Age, married/partnered status

Exclusion Criteria:

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-09-04 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

PRIMARY OUTCOMES:
Communication of genetic test results | 1 Month
  A binary (yes/no) epidemiological item to determine if parental communication of genetic test results occurred to the child.

IPD SHARING:
Plan to Share IPD: No